CLINICAL TRIAL: NCT06347276
Title: De Novo Cerebral Microembolization Associated With Patent Foramen Ovale Closure
Brief Title: Cerebral Microembolization Associated With PFO Closure
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Beijing Anzhen Hospital (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Tibet Autonomous Region People's Hospital (Other); Beijing Tiantan Hospital (Other); Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-RW320-08
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Thrombosis Cardiac; Atrial Septal Defect; Patent Foramen Ovale (PFO)
Keywords: Patent foramen ovale; stroke; migraine; thrombus
MeSH Terms: conditions — Heart Septal Defects, Atrial; Foramen Ovale, Patent; Stroke; Migraine Disorders; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PFO closure: Before PFO closure, all patients will undergo brain DW-MRI. During PFO closure, all patients will undergo right atrial angiography to opacify the PFO, and OCT is used to evaluate the PFO microstructure during angiography while the patient performs the Valsalva maneuver. The presence or absence of in situ thrombus within the PFO will be determined, and thrombus size will be measured. Postoperatively, DW-MRI will be performed 24 hours and one month after the transcatheter closure procedure.
  Interventions: Device: PFO occluder; ASD occluder
- ASD closure: Before ASD closure, all patients will undergo brain DW-MRI. After the transcatheter closure of ASD, DW-MRI will be performed 24 hours and one month postoperatively.
  Interventions: Device: PFO occluder; ASD occluder

INTERVENTIONS:
Device: PFO occluder; ASD occluder — Transcatheter closure of atrial septal defect (ASD) and patent foramen ovale (PFO) All cases will be examined with DW-MRI preoperatively, and DW-MRI will be repeated 24 hours and 4 weeks after the transcatheter closure procedure.

SUMMARY:
This study aims to investigate (1) the de novo cerebral microembolization in patients who undergo transcatheter closure of PFO or ASD, and (2) evaluate the relationship between de novo cerebral microembolization and in situ thrombus within PFO.

DETAILED DESCRIPTION:
Patent foramen ovale (PFO) is prevalent in the general population and it is commonly accepted that PFO is associated with various pathological conditions, including ischemic stroke, transient ischemic attack, migraines, and systemic or coronary embolization. In situ thrombus formation may play a role in patients with PFO-associated stroke or migraines. After transcatheter closure of PFO, peri-interventional cerebral embolic lesions have been detected. This study aims to investigate (1) the de novo cerebral microembolization in patients who undergo transcatheter closure of PFO or ASD, and (2) evaluate the relationship between de novo cerebral microembolization and in situ thrombus within PFO.

ELIGIBILITY:
PFO group

Inclusion Criteria:

1) age 18 to 65 years; 2) documented PFO with medium-to-large shunts (≥ 20 microbubbles by c-TCD at rest or during the Valsalva maneuver); 3) history of embolic stroke (based on brain magnetic resonance imaging within 24 hours after symptom onset) or TIA within 6 months without other identifiable causes; 4) history of migraine for more than one year without other identifiable causes; 5) asymptomatic group: incidental finding of PFO in asymptomatic individuals, and presence of high-risk activities and/or anatomical features related to PFO (high-risk activities were defined as those in which the Valsalva maneuver was performed frequently or those that increased the risk of venous gas formation; and high-risk anatomical features included atrial septal aneurysm and/or curtain pattern on c-TCD).

Exclusion Criteria:

1) presence of any known vascular risk factor, including hypertension, hypercholesterolemia, diabetes mellitus, atrial fibrillation, smoking and obesity; 2) history of embolic stroke or TIA within the past one month; 3) history of deep vein thrombosis or pulmonary embolism; 4) presence of coronary artery disease and carotid artery lesions; 5) presence of coexistent cardiovascular structural malformations or diseases; 6) allergy to contrast medium; 7) refusal to participate.

ASD group

Inclusion Criteria:

1) age 18 to 65 years; 2) secundum ASD size 10 to 20 mm, with sufficient surrounding rims, except the aortic rim; 3) right heart catheterization: resting SPAP < 50 mm Hg, Qp/Qs ≥ 1.5 and PVR < 5 WU.

Exclusion Criteria:

1) presence of any known vascular risk factor, including hypertension, hypercholesterolemia, diabetes mellitus, atrial fibrillation, smoking and obesity; 2) associated with other cardiac abnormalities or diseases; 3) resting SPAP ≥50 mm Hg and resting PVR ≥5 Wood units;4) primum or sinus venosus type ASD; 5) presence of intracardiac thrombi, permanent contraindications to platelet therapy, and allergic reaction to nickel.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, there are two groups of the patients who will undergo transcatheter closure. (1) PFO patients (n=600); (2) ASD patients (n=200). Before transcatheter closure, all patients will undergo brain DW-MRI. After the transcatheter closure, DW-MRI will be performed 24 hours and 4 weeks postoperatively. In addition, the presence or absence of in situ thrombus within the PFO will be determined in patients with PFO.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
De novo cerebral microembolization | 24 hours to 4 weeks after closure of PFO/ASD
  cerebral microembolization with diffusion-weighted magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Chaowu Yan, PhD MD, Principal Investigator — Cardiovascular Institute and Fuwai Hospital
Locations (1):
- Chaowu Yan, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
he data that support the findings of this study are available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Yan C, Li H, Wang C, Yu H, Guo T, Wan L, Yundan P, Wang L, Fang W. Frequency and Size of In Situ Thrombus Within Patent Foramen Ovale. Stroke. 2023 May;54(5):1205-1213. doi: 10.1161/STROKEAHA.122.041524. Epub 2023 Mar 9. PMID 36891906
- [Background] Yan C, Li H. Preliminary Investigation of In situ Thrombus Within Patent Foramen Ovale in Patients With and Without Stroke. JAMA. 2021 May 25;325(20):2116-2118. doi: 10.1001/jama.2021.4359. PMID 34032839